CLINICAL TRIAL: NCT02825121
Title: Evaluation of Monitoring Neuromuscular Blockade the Flexor Hallucis Compared to the Adductor Pollicis
Acronym: CurHaTOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CURHATOF
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2016-10

CONDITIONS: Observation of Neuromuscular Block; Flexor Hallucis; Adductor Pollicis

ARMS (1):
- Monitoring Neuromuscular Blockade (Experimental): Monitoring Neuromuscular Blockade the Flexor Hallucis and adductor of the thumb.
  Interventions: Device: Monitoring Neuromuscular Blockade the Flexor Hallucis; Device: Monitoring Neuromuscular Blockade adductor of the thumb.

INTERVENTIONS:
Device: Monitoring Neuromuscular Blockade the Flexor Hallucis
Device: Monitoring Neuromuscular Blockade adductor of the thumb.

SUMMARY:
Current guidelines recommend monitoring of neuromuscular blockade at the adductor pollicis by stimulation of the ulnar nerve at the wrist.

However, in certain situations (laparoscopic surgery, cranial surgery or surgical comfort, arterial catheterization), it is impossible to access the patient's wrists, delaying monitoring, antagonizing the neuromuscular block, the emergence from anesthesia and patient extubation , leading in some cases to single injections lack of control of the reversal of the patient.

To overcome these technical difficulties, a group nerve / muscle looks interesting and often easily accessible to the anesthesiologist.

The stimulation of the posterior tibial nerve can observe a response to the flexor hallucis brevis muscle and allows quick access to monitoring the reversal before the end of the intervention.

The primary outcome was to compare the speed of recovery from neuromuscular block flexor hallux versus that of the adductor pollicis.

The secondary objective was to compare the speed of installation of deep neuromuscular block flexor hallucis versus that of the adductor pollicis.

This is a prospective, exploratory, uncontrolled, single-center for routine care.

Are included all aged patients over 18 years, ASA I or II, without guardianship, having no known allergy to Atracurium, without neuromyopathy known, emergency surgery or full stomach, predictable difficult intubation .

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* Any elective surgery with single or multiple injection Atracurium for which hand and foot are accessible at the same time.
* ASA I or II patients
* free subject, without guardianship or subordination
* No opposition given by the patient after information

Exclusion Criteria:

* under 18 years
* known neuromyopathy
* Diabetics
* Emergency surgery and a full stomach
* predictable difficult intubation
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Time of occurrence of a T4 / T1 ratio> 0.90 in the train of four flexor hallucis | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers Universitary Hospital, Poitiers, France

REFERENCES:
- [Derived] Le Merrer M, Frasca D, Dupuis M, Debaene B, Boisson M. A comparison between the flexor hallucis brevis and adductor pollicis muscles in atracurium-induced neuromuscular blockade using acceleromyography: A prospective observational study. Eur J Anaesthesiol. 2020 Jan;37(1):38-43. doi: 10.1097/EJA.0000000000001090. PMID 31592900